CLINICAL TRIAL: NCT02903524
Title: The Efficacy and Safety of Doxorubicin Hydrochloride Liposome Injection Plus Cyclophosphamide Compared to Pirarubicin Plus Cyclophosphamide as Neoadjuvant Chemotherapy in Locally Advanced Breast Cancer ：a Randomised Multicentre, Open-label Trial
Brief Title: Doxorubicin Hydrochloride Liposome Injection Combination With Cyclophosphamide vs Pirarubicin Combination With Cyclophosphamide in Patients With Locally Advanced Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-BC-03
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; pirarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Active Comparator): Pirarubicin combination with cyclophosphamide,4 cycles (each cycle is 21days) of chemotherapy
  Interventions: Drug: pirarubicin and cyclophosphamide
- Experimental group (Experimental): Doxorubicin Hydrochloride Liposome Injection combination with cyclophosphamide, 4 cycles (each cycle is 21 days) of chemotherapy
  Interventions: Drug: Doxorubicin Hydrochloride Liposome injection and cyclophosphamide

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride Liposome injection and cyclophosphamide
  Arms: Experimental group
Drug: pirarubicin and cyclophosphamide
  Arms: control group

SUMMARY:
Evaluate the efficacy and safety of Doxorubicin Hydrochloride Liposome Injection Plus Cyclophosphamide Compared to Pirarubicin Plus Cyclophosphamide as Neoadjuvant Chemotherapy in Locally Advanced Breast Cancer Patients

ELIGIBILITY:
Inclusion Criteria:

* Female patients with age between 18 and 70 years.
* Newly diagnosed breast cancer, stages IIb-IIIc.
* KPS performance status≥70.
* Measurable disease according to RECIST version 1.1.
* Normal cardiac function confirmed by baseline left ventricular ejection fraction (LVEF)≥50%.
* Adequate bone marrow reserve (WBC≥4.0×10(9)/L, neutrophils≥2.0×10(9)/L, platelets≥100×10(9)/L,and hemoglobin≥90g/L).
* Adequate hepatic and renal function.
* AST and ALT ≤ 2×institutional upper limit of normal；alkaline phosphatase ≤ 2×institutional upper limit of normal；bilirubin ≤ institutional upper limit of normal.
* Serum creatinine≥44 µmol/L and ≤133 µmol/L.
* Written informed consent are acquired.
* Not in pregnancy or the pregnancy tests of females is negative.

Exclusion Criteria:

* Severe heart failure (NYHA grade II or higher).
* Active and uncontrolled severe infection.
* Have accepted any other anti-tumor drug within 30 days before the first dose or
* received radiation treatment.
* Other situations that investigators consider as contra-indication for this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
pathological complete response | until the completion of 4 cycles (each cycle is 21 days) of chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China